CLINICAL TRIAL: NCT05982327
Title: Assessment of Operative Management of Scapular Fractures in Level 1 Trauma Center
Brief Title: Operative Management of Scapular Fractures
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Elbadry Mahmoud Ahmed, Assuit lecturer, Assiut University
Other Study IDs: Scapular fractures
Record Dates: First submitted 2023-07-19; First posted 2023-08-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Scapular Fracture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ORIF — fixation of scapular fractures by plate and screws

SUMMARY:
Assessment of functional outcome of operative management of scapular fractures through Arabic version DASH score

DETAILED DESCRIPTION:
Scapular fractures are rare, accounting less than1% all fractures. 3-5%all fractures of shoulder girdle, however very serious because 80-90% due to high energy trauma such as Motor car accidents or Fall from height. It can be associated with life-threatening injuries such as thoraco-scapular dissociation and vascular injury as subclavian and axillary vessels and brachial plexus injuries.So morbidity and mortality reports are relatively high.It can be diagnosed by X ray and computed tomography scan (CT scan) that play important role to discover scapular fractures and associated injuries ,and to guide clinical decision such as approaches and other surgical interventions.Most of scapular fractures are managed conservatively by Immbolization in sling .literature stated that conservative management of scapular body fractures and scapular neck fractures displaced less than 10 mm have satisfactory outcome and operative management suitable for displaced glenoid fossa fractures and scapular neck fractures more than 10 mm and associated with better functional outcome.Others stated that conservative management with highly displaced scapular body and neck fractures are associated with satisfactory long -term functional outcome with minor loss of motion and strength.

So standard treatment of scapular fracture is still controversial and there is no clear guidelines about management of scapular fractures.

In Investigators hypothesis, Operative management of scapular fractures is better choice due to better functional outcome, early rehabilitation ,high union rate and less complications. Investigators will try to answer this question ''What is the effect of operative management of scapular fractures on functional outcome?''

ELIGIBILITY:
Inclusion Criteria:

* 1.All patient presented with scapular fractures more than 18 years old involving body, neck and glenoid 2.Intraarticular glenoid fractures with step-off >4 mm 3.>20% of the joint is involved and Fragment large enough to be hold by lag screw.

Exclusion Criteria:

1- Low demanded patients:Age >65 yrs . 2.Scapular fractures of acromion and coracoid process and Osteoporotic fractures .

3.Scapular fractures associated with brain injuries cervical spine injuries and brachial plexus injuries.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patients who meets the inclusion criteria and agrees to be involved in our study will do:
  1. Preoperative assessment:
     1. Examination : Neurological and Vascular examination
     2. Imaging:
        * Plain X- ray (True AP - Scapula Y view ) and Plain X-ray (True AP )of contralateral side Measurement of Glenopolar angle (GPA)
        * CT scan
  2. Intra-operative assessment:
     a. Selection of approach. b.Postion C.Type of osteosynthesis d. Blood loss e. Radiation exposure.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-05 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of functional outcome | 6 week
  Arabic version DASH score

SECONDARY OUTCOMES:
Range of motion | Six months
  Goniometer
Strength of shoulder muscle | Six months
  Handheld dynamometer
Union rate | Six months
  X ray-CT

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elbadry Mahmoud, Resident, Principal Investigator — Assiut University; Aly Mohamadean, Prof Dr, Study Director — Assiut University; Mahmoud Badran, Ass.prof, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ideberg R, Grevsten S, Larsson S. Epidemiology of scapular fractures. Incidence and classification of 338 fractures. Acta Orthop Scand. 1995 Oct;66(5):395-7. doi: 10.3109/17453679508995571. PMID 7484114
- [Result] Voleti PB, Namdari S, Mehta S. Fractures of the scapula. Adv Orthop. 2012;2012:903850. doi: 10.1155/2012/903850. Epub 2012 Nov 20. PMID 23209916
- [Result] McGahan JP, Rab GT, Dublin A. Fractures of the scapula. J Trauma. 1980 Oct;20(10):880-3. doi: 10.1097/00005373-198010000-00011. PMID 6252325
- [Result] Zelle BA, Pape HC, Gerich TG, Garapati R, Ceylan B, Krettek C. Functional outcome following scapulothoracic dissociation. J Bone Joint Surg Am. 2004 Jan;86(1):2-8. doi: 10.2106/00004623-200401000-00002. PMID 14711938
- [Result] Brown CV, Velmahos G, Wang D, Kennedy S, Demetriades D, Rhee P. Association of scapular fractures and blunt thoracic aortic injury: fact or fiction? Am Surg. 2005 Jan;71(1):54-7. PMID 15757058
- [Result] Lantry JM, Roberts CS, Giannoudis PV. Operative treatment of scapular fractures: a systematic review. Injury. 2008 Mar;39(3):271-83. doi: 10.1016/j.injury.2007.06.018. Epub 2007 Oct 4. PMID 17919636
- [Result] Kannan S, Singh HP, Pandey R. A systematic review of management of scapular fractures. Acta Orthop Belg. 2018 Dec;84(4):497-508. PMID 30879456
- [Result] Mayo KA, Benirschke SK, Mast JW. Displaced fractures of the glenoid fossa. Results of open reduction and internal fixation. Clin Orthop Relat Res. 1998 Feb;(347):122-30. PMID 9520882